CLINICAL TRIAL: NCT00461357
Title: Outcome After Renal Transplantation of a Randomized Prospective Trial in the Eurotransplant Senior Program
Brief Title: Sirolimus Based Immunosuppression for Patients Undergoing Kidney Transplantation in the Eurotransplant Senior Program
Acronym: ESP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Other Study IDs: NTX-OFO-01
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Last update posted 2007-04-18 (Estimated); Status verified 2007-04

CONDITIONS: Kidney Function After Transplantation; Outcome After Kidney Transplantation
Keywords: Old for Old; Eurotransplant Senior Program; Glomerular Filtration Rate

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Eurotransplant Senior Program (ESP) started in 1999 with local allocation of kidneys from deceased donors elder than 65 years to recipients elder than 65 years. The requirements for immunosuppression in this group of patients are high due to the large amount of comorbidities.

This prospective randomized trial compared the standard immunosuppressive protocol based on cyclosporine A (CyA) used at our center within the ESP, to a calcineurin inhibitor-free protocol based on sirolimus (SRL).

The aim of this study is to investigate the effect of a CNI-free therapy on the function of elderly kidneys 6 months post transplantation, measured by GFR.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of the Eurotransplant Senior Program
* negative cytotoxic crossmatch
* signed informed consent

Exclusion Criteria:

* High sensitized recipients (PRA > 40%)
* Non heart Beating Donor
* Hyperlipidemia
* Leucocytopenia (< 3000/mm3)
* Thrombocytopenia (< 75000/mm3)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48
Dates: Start 2003-01; Study Completion 2007-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ferdinand Muehlbacher, MD Professor, Principal Investigator — Medical University of Vienna; Department of Transplantation